CLINICAL TRIAL: NCT05334524
Title: Effects of Kinesiotaping With and Without Combined Chain Exercises on Pain, Range of Motion and Quality of Life in Patients With Knee Osteoarthritis
Brief Title: Kinesiotaping With and Without Combined Chain Exercises in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0132 Sobia
Record Dates: First submitted 2022-04-02; First posted 2022-04-19 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Kinesiotaping; Combined chain exercises; Pain; ROM; quality of life
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesiotaping with combined chain exercises (Active Comparator): 3 Kinesiotape strips will be applied: 2 "Y-strips" with a length of approximately 20 cm and an anchor of 2 cm and a single longitudinal section (1 "I-strip"). Tails of the quadriceps strip were applied to the patella, wrapping the patella medially and laterally with 25% tension and the (I-strip) will be applied with 75% tension.
  Combined chain exercises will apply with 10 secs hold with 10 repetitions which will include quadriceps setting, SLR, full arc extension, cycling in the air, wall slides and step-up and step-down exercises.
  Interventions: Other: kinesiotaping with combined chain exercises; Other: kinesiotaping
- kinesiotaping (Active Comparator): 3 Kinesiotape strips will be applied: 2 "Y-strips" with a length of approximately 20 cm and an anchor of 2 cm and a single longitudinal section (1 "I-strip"). Tails of the quadriceps strip were applied to the patella, wrapping the patella medially and laterally with 25% tension and the (I-strip) will be applied with 75% tension.
  Interventions: Other: kinesiotaping

INTERVENTIONS:
Other: kinesiotaping with combined chain exercises — 3 Kinesiotape strips will be applied: 2 "Y-strips" with a length of approximately 20 cm and an anchor of 2 cm and a single longitudinal section (1 "I-strip"). Tails of the quadriceps strip were applied to the patella, wrapping the patella medially and laterally with 25% tension and the (I-strip) will be applied with 75% tension.
  Combined chain exercises will apply with 10 secs hold with 10 repetitions which will include quadriceps setting, SLR, full arc extension, cycling in the air, wall slides and step-up and step-down exercises
  Arms: kinesiotaping with combined chain exercises
Other: kinesiotaping — 3 Kinesiotape strips will be applied: 2 "Y-strips" with a length of approximately 20 cm and an anchor of 2 cm and a single longitudinal section (1 "I-strip"). Tails of the quadriceps strip were applied to the patella, wrapping the patella medially and laterally with 25% tension and the (I-strip) will be applied with 75% tension

SUMMARY:
Knee osteoarthritis is a major public health issue because it causes chronic pain, reduces physical function and diminishes quality of life. Aging of the population and increased global prevalence of obesity are anticipated to dramatically increase the prevalence of knee osteoarthritis. Knee osteoarthritis is characterized by complex multifactorial joint pathology and is the most common form of joint disorder in the world. Chronic knee osteoarthritis leads to marked weakening of the quadriceps femoris muscle, which is the extensor and stabilizer of the knee and atrophy of this muscle result knee pain and functional impairment. Quadriceps muscle weakness and atrophy have been reported to contribute to functional impairment and pain in patients with knee osteoarthritis and quadriceps strengthening can be achieved through open kinetic chain exercises and close kinetic chain exercises. Close kinetic chain exercises are modeled as, in which a movement in a joint simultaneously produces movements in other joints of the extremity. Open kinetic chain exercises and close kinetic chain exercises form the combined chain exercises. Kinesiotaping with these exercises to improve the patients suffering with knee osteoarthritis. The aim of this study will be to compare the effects of kinesiotaping as an adjunct to combined chain exercises compared with only kinesiotaping on pain, range of motion and quality of life in the management of individuals with knee osteoarthritis.

This study will be randomized control trial. Patients will be recruited into two groups by simple random assignment. Non probability consecutive sampling technique will be used. Data will be collected from patients of grade 2 knee osteoarthritis patients by using NPRS for pain, Goniometer for ROM and SF-36 for quality of life will be used before and immediate after the treatment. Those who will meet the inclusion criteria will be recruited. Group 1 will be treated with kinesiotaping and combined chain exercises and the Group 2 will be treated with only kinesiotaping on knee OA patients. Total intervention will be given for four weeks for three sessions per week.The subject attended physical therapy and kinesiotaping will assess for pain, range of motion and quality of life at baseline and after 4 week of intervention. After collecting data from defined study setting, data will be entered and analyzed by using Statistical Package for the Social Sciences (SPSS) for Windows software, version 25.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients.
* Patients age between 40 years- 60years.
* Patients with Grade II knee osteoarthritis.

Exclusion Criteria:

* Patients with allergic reaction to tape or any skin problems
* Patients with history of injection at the knee.
* Patients with surgical intervention at the knee

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
NPRS | 4th week
  used for pain measurement, It is a uni-dimensional 11 point scale (0-10) with measure of pain intensity with High test-retest reliability of r = 0.96 and validity correlations range from 0.86 to 0.95 (7).
Goniometry | 4th week
  It is a device that measures an angle or permits the rotation of an object to a definite position
SF-36 Questionnaire | 4th week
  For quality of life SF-36 questionnaire is used. The questionnaire consists of 36 items on physical and social functioning and has 8 domains. The total score ranges from 0 to 100, with higher scores indicating better quality of life and lower scores indicating the worse quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Hina Gul, t-DPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaya Mutlu E, Mustafaoglu R, Birinci T, Razak Ozdincler A. Does Kinesio Taping of the Knee Improve Pain and Functionality in Patients with Knee Osteoarthritis?: A Randomized Controlled Clinical Trial. Am J Phys Med Rehabil. 2017 Jan;96(1):25-33. doi: 10.1097/PHM.0000000000000520. PMID 27149590
- [Background] Olagbegi OM, Adegoke BOA, Odole AC. Effectiveness of combined chain exercises on pain and function in patients with knee osteoarthritis. Bangladesh Journal of Medical Science. 2016;15(2):178-88.
- [Background] Danazumi MS, Ibrahim SU, Yakasai AM, Dermody G, Bello B, Kaka B. A Comparison Between the Effect of Combined Chain Exercises Plus Kinesio Taping With Combined Chain Exercises Alone in Knee Osteoarthritis: A Randomized Clinical Trial. Am J Phys Med Rehabil. 2021 Nov 1;100(11):1070-1077. doi: 10.1097/PHM.0000000000001705. PMID 33496439
- [Background] Rahlf AL, Braumann KM, Zech A. Kinesio Taping Improves Perceptions of Pain and Function of Patients With Knee Osteoarthritis: A Randomized, Controlled Trial. J Sport Rehabil. 2019 Jul 1;28(5):481-487. doi: 10.1123/jsr.2017-0306. Epub 2018 Dec 12. PMID 29466081
- [Background] Abolhasani M, Halabchi F, Afsharnia E, Moradi V, Ingle L, Shariat A, Hakakzadeh A. Effects of kinesiotaping on knee osteoarthritis: a literature review. J Exerc Rehabil. 2019 Aug 28;15(4):498-503. doi: 10.12965/jer.1938364.182. eCollection 2019 Aug. PMID 31523668
- [Background] Ye W, Jia C, Jiang J, Liang Q, He C. Effectiveness of Elastic Taping in Patients With Knee Osteoarthritis: A Systematic Review and Meta-Analysis. Am J Phys Med Rehabil. 2020 Jun;99(6):495-503. doi: 10.1097/PHM.0000000000001361. PMID 31851010
- [Background] Olagbegi OM, Adegoke BO, Odole AC. Effectiveness of three modes of kinetic-chain exercises on quadriceps muscle strength and thigh girth among individuals with knee osteoarthritis. Arch Physiother. 2017 Jul 19;7:9. doi: 10.1186/s40945-017-0036-6. eCollection 2017. PMID 29340203